CLINICAL TRIAL: NCT04161742
Title: Evaluation of the Clinical Utility of Electrical Impedance Spectroscopy in Normal Clinical Practice at Hospital Setting
Brief Title: Clinical Utility of Electrical Impedance Spectroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SciBase AB (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FG-001
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Focus of Study: Patients With Suspicion of Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Nevisense — Nevisense measures electrical impedance of skin lesions and provides an output called the electrical impedance spectroscopy (EIS) score

SUMMARY:
The purpose of this clinical study is to evaluate the clinical utility of the Nevisense in normal clinical practice, i.e. the potential effect of implementing Nevisense in clinical decision making (Human vs Human & Machine) based on Nevisense measurement at time of biopsy decision.

DETAILED DESCRIPTION:
This is a multi-center, prospective, blinded clinical study designed to evaluate clinical utility of Nevisense in normal clinical practice, i.e. the potential effect of implementing Nevisense in clinical decision making (Human vs Human & Machine) based on Nevisense measurement after biopsy decision. The study enrollment will continue until minimum of 180 subjects are enrolled in the study. Up to 3 US university/hospital investigational sites will participate in this study. Biopsying clinician or the investigators from the clinical practices of physicians participating in the study will perform the patient and lesion assessment for biopsy as standard of care at the clinic.

Study subjects will be recruited from the clinical practices of physicians participating as investigators in this study. Biopsying clinicians provide their assessment to whether s/he would have sent the lesion(s) for biopsy had s/he known the EIS information beforehand . Thereafter an evaluation of the suspicious lesion with the Nevisense will be performed followed by a biopsy of the lesion. The biopsied lesion will be subjected to histological analysis.

ELIGIBILITY:
Inclusion Criteria:

* The lesion(s) meet criteria for Nevisense evaluation.
* Lesions that present with unclear clinical presentation to allow for clinical diagnosis of benign or minimally dysplastic nevus (nevi) -Thus, necessitating a biopsy.
* Lesions within Nevisense indication for use: Nevisense is indicated for use on cutaneous lesions with one or more clinical or historical characteristics of melanoma, when a dermatologist chooses to obtain additional information when considering biopsy. Nevisense should not be used on clinically obvious melanoma. The Nevisense result is one element of the overall clinical assessment. The output of Nevisense should be used in combination with clinical and historical signs of melanoma to obtain additional information prior to a decision to biopsy. Nevisense is indicated only for use on:

  * primary skin lesions with a diameter between 2 mm and 20 mm;
  * lesions that are accessible by the Nevisense probe;
  * lesions where the skin is intact (i.e. non-ulcerated or non-bleeding lesions);
  * lesions that do not contain a scar or fibrosis consistent with previous trauma;
  * lesions not located in areas of psoriasis, eczema, acute sunburn or similar skin conditions;
  * lesions not in hair-covered areas;
  * lesions which do not contain foreign matter;
  * lesions not on special anatomic sites (i.e. not for use on acral skin, genitalia, eyes, mucosal areas).

Exclusion Criteria:

* Subjects who fail to provide informed consent
* Study subjects with underlying medical disease which may alter ability to diagnose clinically or inhibit Nevisense from collecting data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Number needed to biopsy | 1 day
  The primary study outcome is the number needed to biopsy to detect a single melanoma case.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ferris, MD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malvehy J, Hauschild A, Curiel-Lewandrowski C, Mohr P, Hofmann-Wellenhof R, Motley R, Berking C, Grossman D, Paoli J, Loquai C, Olah J, Reinhold U, Wenger H, Dirschka T, Davis S, Henderson C, Rabinovitz H, Welzel J, Schadendorf D, Birgersson U. Clinical performance of the Nevisense system in cutaneous melanoma detection: an international, multicentre, prospective and blinded clinical trial on efficacy and safety. Br J Dermatol. 2014 Nov;171(5):1099-107. doi: 10.1111/bjd.13121. Epub 2014 Oct 19. PMID 24841846
- [Background] Rocha L, Menzies SW, Lo S, Avramidis M, Khoury R, Jackett L, Guitera P. Analysis of an electrical impedance spectroscopy system in short-term digital dermoscopy imaging of melanocytic lesions. Br J Dermatol. 2017 Nov;177(5):1432-1438. doi: 10.1111/bjd.15595. Epub 2017 Oct 11. PMID 28421597